CLINICAL TRIAL: NCT04894305
Title: A Phase 1, Randomized, Observer-blind Study to Compare the Safety, Reactogenicity, and Immunogenicity of Ad26.COV2.S at a Single Dose of 5*10^10 vp in 2 Different Volumes in Healthy Adults
Brief Title: A Study of Ad26.COV2.S in Healthy Adults (COVID-19)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Vaccines & Prevention B.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CR109013; 2021-001374-30 (EudraCT Number); VAC31518COV1003 (Other: Janssen Vaccines & Prevention B.V.)
Expanded Access: NCT04817657 (No longer available)
Record Dates: First submitted 2021-05-18; First posted 2021-05-20 (Actual); Last update posted 2021-12-22 (Actual); Status verified 2021-12

CONDITIONS: Healthy
MeSH Terms: interventions — Ad26COVS1

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group 1 (Test Group): Ad26.COV2.S (0.3 mL) (Experimental): Participants will receive single dose Ad26.COV2.S 0.3 milliliter (mL) intramuscular (IM) injection on Day 1 in test group.
  Interventions: Biological: Ad26.COV2.S
- Group 2 (Reference Group): Ad26.COV2.S (0.5 mL) (Active Comparator): Participants will receive single dose Ad26.COV2.S 0.5 mL IM injection on Day 1 in reference group.
  Interventions: Biological: Ad26.COV2.S

INTERVENTIONS:
Biological: Ad26.COV2.S — Ad26.COV2.S will be administered as IM injection.
  Other Names: JNJ-78436735, VAC31518

SUMMARY:
The purpose of this study is to assess the safety and reactogenicity of Ad26.COV2.S (0.3 milliliter [mL] versus 0.5 mL) and to demonstrate non-inferiority (NI) of Ad26.COV2.S (0.3 mL versus 0.5 mL), 28 days after vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Participant must sign an informed consent form (ICF) indicating that he or she understands the purpose, procedures and potential risks and benefits of the study, and is willing to participate in the study
* Participant must be healthy, in the investigator's clinical judgment, as confirmed by medical history, physical examination, and vital signs performed at screening. Participant may have underlying illnesses, as long as the symptoms and signs are medically controlled and not considered to be comorbidities related to an increased risk of severe coronavirus disease-2019 (COVID-19), except for smoking, which is allowed. If on medication for a condition, the medication dose must have been stable for at least 12 weeks preceding vaccination and expected to remain stable for the duration of the study
* All participants of childbearing potential must: a) have a negative highly sensitive urine pregnancy test at screening; b) have a negative highly sensitive urine pregnancy test immediately on the day of and prior to study vaccine administration
* Participant agrees to not donate bone marrow, blood, and blood products from the first study vaccine administration until 3 months after receiving the study vaccine
* Participant must be willing to provide verifiable identification, has means to be contacted and to contact the investigator during the study

Exclusion Criteria:

* Participant has a history of malignancy within 5 years before screening (exceptions are squamous and basal cell carcinomas of the skin and carcinoma in situ of the cervix, or malignancy, which is considered cured with minimal risk of recurrence)
* Participant has a known or suspected allergy or history of anaphylaxis or other serious adverse reactions to vaccines or their excipients (including specifically the excipients of the study vaccine)
* Participant has a history of any neurological disorders or seizures including Guillain-barre syndrome, with the exception of febrile seizures during childhood
* Participant has a history of chronic urticaria (recurrent hives), eczema or adult atopic dermatitis
* Participant received treatment with immunoglobulins in the 3 months or exogenous blood products (autologous blood transfusions are not exclusionary) in the 4 months before the planned administration of the study vaccine or has any plans to receive such treatment during the study
* Upper limit of body mass index (BMI) range should not be considered in participants with comorbidities that are or might be associated with an increased risk of progression to severe COVID-19. Participants may have hypertension of mild severity, as long as it is stable and medically controlled as defined by no change in medication over the past 6 months (except for issues of tolerability or use of similar drug with same mechanism of action, example, thiazides, beta blockers, alpha blockers at the same effective dose)
* Participant who is an employee of the sponsor, investigator or study site with direct involvement in the proposed study or other studies under the direction of that investigator or study site, including the family members of those employees or the investigator

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 380 (Actual)
Dates: Start 2021-05-25 (Actual); Primary Completion 2021-12-08 (Actual); Study Completion 2021-12-08 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Solicited Local Adverse Events (AEs) for 7 Days After Vaccination | Day 8 (7 days after vaccination)
  An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Solicited local AEs are pre-defined local (at the injection site) AEs. Participants will be asked to note in the diary occurrences of injection site pain/tenderness, erythema and swelling at the study vaccine injection site daily for 7 days post vaccination (day of vaccination and the subsequent 7 days).
Number of Participants with Solicited Systemic AEs for 7 Days After Vaccination | Day 8 (7 days after vaccination)
  Number of participants with solicited systemic AEs will be reported. Participants will be instructed on how to record daily temperature using a thermometer and also instructed to note signs and symptoms in the diary on a daily basis for 7 days after vaccination. Solicited systemic AEs are fatigue, headache, nausea, and myalgia.
Number of Participants with Unsolicited AEs for 28 Days After Vaccination | Day 29 (28 days after vaccination)
  Number of participants with unsolicited AEs will be reported. Unsolicited AEs are all AEs for which the participant is not specifically questioned in the participant diary.
Number of Participants with AEs Leading to Study Discontinuation | Up to 6 months
  Number of participants with AEs leading to study discontinuation will be reported.
Number of Participants with Serious Adverse Events (SAEs) | Up to 6 months
  A SAE is any untoward medical occurrence that at any dose: results in death; is life-threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect; is a suspected transmission of any infectious agent via a medicinal product; is medically important.
Number of Participants with Adverse Events of Special Interests (AESIs) | Up to 6 months
  Number of participants with AESIs will be reported. AESIs are significant AEs that are judged to be of special interest because of clinical importance, known or suspected class effects, or based on nonclinical signals. Thrombosis with Thrombocytopenia Syndrome (TTS), a syndrome characterized by a combination of both a thrombotic event and thrombocytopenia, is considered to be an AESI in this study. A suspected TTS case is defined as: Thrombotic events: suspected deep vessel venous or arterial thrombotic events; Thrombocytopenia, defined as platelet count below 150,000/micro liter.
S Enzyme-linked Immunosorbent Assay (S-ELISA) Geometric Mean Concentrations (GMCs) 28 Days After Vaccination | Day 29 (28 days after vaccination)
  Non-inferiority (NI) will be assessed in terms of humoral immune response expressed by the GMCs of S-ELISA.

SECONDARY OUTCOMES:
Severe Acute Respiratory Syndrome Coronavirus(-2) (SARS-CoV-2) S Protein Binding Antibody Concentrations as Measured by S-ELISA | Up to 6 months
  SARS-CoV-2 S protein binding antibody concentrations as measured by S-ELISA will be reported.
Serological Response to Vaccination as Measured by Virus Neutralization Assay (VNA) Titers | Up to 6 months
  Serological response to vaccination, as measured by VNA titers will be reported.
Geometric Mean Titers (GMTs) of Antibody | Up to 6 months
  GMTs of antibody will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Vaccines & Prevention B.V. Clinical Trial, Study Director — Janssen Vaccines & Prevention B.V.
Locations (1):
- PRA Health Sciences, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency